CLINICAL TRIAL: NCT05638061
Title: The Effect of Food Sources of Soy Protein on Blood Pressure: A Systematic Review and Meta-Analysis of Randomized Controlled Trials
Brief Title: SRMA of the Effect of Soy Protein on Blood Pressure
Status: Active, not recruiting | Type: Observational
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, John Sievenpiper, Associate Professor, University of Toronto
Other Study IDs: CIHR - Soy and BP
Record Dates: First submitted 2022-11-10; First posted 2022-12-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Blood Pressure; Cardiovascular Diseases
Keywords: systolic blood pressure; diastolic blood pressure; systematic review; meta-analysis; randomized controlled trial
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Soybean Proteins

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Soy protein — Soy foods or isolated soy protein
  Other Names: Soya, soybean, soy bean, soya bean

SUMMARY:
Hypertension is one of the leading risk factors for death and significantly increases the risk for cardiovascular (CVD), brain and kidney diseases. It is also one of the leading modifiable risk factors for CVD, which also plays a significant role in the global burden of death and disease. Dietary guidelines for blood pressure management and hypertension emphasize fruits and vegetables, plant-based proteins and foods low in saturated fat. With the growing interest in plant-based alternatives and plant-based diets, there is a need to clarify their benefits on blood pressure. Soy protein is a complete protein and is the only plant-based beverage alternative that is comparable to dairy milk. There are mixed findings on the effects of soy on blood pressure due to differences in study design and subjects. To better address this question and inform public health guidelines the investigators will conduct a systematic review and meta-analysis of randomized controlled trials of the effect of soy protein on reducing blood pressure in individuals with and without hypertension.

DETAILED DESCRIPTION:
RATIONALE: Hypertension is one of the leading risk factors for death and significantly increases the risk for cardiovascular disease (CVD), brain and kidney diseases. It is also one of the leading modifiable risk factors for CVD. Dietary guidelines for blood pressure management and hypertension emphasize fruits and vegetables, plant-based proteins and foods low in saturated fat. With the growing interest in plant-based alternatives and plant-based diets, there is a need to clarify their benefits on blood pressure. Soy protein is a complete protein and is the only plant-based beverage alternative that is comparable to dairy milk. There are mixed findings on the effects of soy on blood pressure due to differences in study design and subjects. To better address this question and inform public health guidelines the investigators will conduct a systematic review and meta-analysis of randomized controlled trials of the effect of soy protein on reducing blood pressure in individuals with and without hypertension.

OBJECTIVES: To conduct a systematic review of the effect of soy protein by food source on systolic (SBP) and diastolic (DBP) blood pressure in individuals with and without hypertension and assess the certainty of the evidence using the Grading of Recommendations Assessment Development and Evaluation (GRADE) system.

DESIGN: The systematic review and meta-analyses will be conducted according to the Cochrane Handbook for Systematic Reviews of Interventions and reported according to the Preferred Reporting items for Systematic Reviews and Meta-Analyses (PRISMA).

DATA SOURCES: Medline, Embase, and The Cochrane Central Register of Controlled Trials (Clinical Trials; CENTRAL) will be searched using appropriate search terms supplemented by manual searches of references of included studies.

STUDY SELECTION: Randomized controlled trials of ≥3-weeks assessing the effect of soy protein food sources compared with a suitable non-soy-containing control group on blood pressure will be included.

DATA EXTRACTION: Two or more investigators will independently extract relevant data. Authors will be contacted for additional information and any missing data will be computed/imputed using standard formulae.

RISK OF BIAS: Two or more investigators will independently assess risk of bias using the Cochrane Risk of Bias Tool. All disagreements will be resolved by consensus.

OUTCOMES: The primary outcomes will be SBP and DBP.

DATA SYNTHESIS: Data will be pooled using the Generic Inverse Variance method for each outcome. Random effects models will be used even in the absence of statistically significant between-study heterogeneity, as they yield more conservative summary effect estimates in the presence of residual heterogeneity. Fixed-effects models will only be used where there is <5 included studies. Paired analyses will be applied for crossover design trials. Heterogeneity will be assessed (Cochran Q statistic) and quantified (I2 statistic). Sources of heterogeneity will be explored (if there are >=10 trial comparisons) by sensitivity analyses and a priori subgroup analyses (dose, soy protein food source, comparator, follow-up, baseline levels, design, age, health status, funding and risk of bias). Meta-regression analyses will assess the significance of categorical and continuous subgroups analyses. Publication bias will be assessed (if there are >=10 trial comparisons) by inspection of funnel plots and the Egger and Begg tests. Adjustment for evidence of funnel plot asymmetry or small study effects will be conducted by the Duval and Tweedie trim-and-fill method.

GRADE ASSESSMENT. To assess the certainty of the evidence, the investigators will use the GRADE system, an evidence-based grading system adopted by >100 organizations (http://www.gradeworkinggroup.org/). It grades the evidence as high, moderate, low or very low quality based on the study design and a series of downgrades (risk of bias, imprecision, inconsistency, indirectness, publication bias) and upgrades (large magnitude of the effect, dose-response gradient, and attenuation by confounding). The investigators will follow the GRADE handbook (https://gdt.gradepro.org/app/handbook/handbook.html) and use the GRADEpro GDT (gradepro.org) software.

SIGNIFICANCE: The proposed evidence synthesis will assess the role of different food sources of soy protein for blood pressure management, increasing the evidence-base for health claims and guidelines development and improving health outcomes, by educating healthcare providers and patients, stimulating industry innovation, and guiding future research design.

ELIGIBILITY:
Inclusion Criteria:

* Randomized Controlled Trials
* Soy intervention
* Non-soy comparator
* Intervention duration >3 weeks
* Data for >1 Outcome

Exclusion Criteria:

* Observational Studies
* Non-Human Studies
* Lack of Suitable Comparator (i.e. soy-containing, equally matched doses)
* Multimodal interventions
* RCTs with participants < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with or without high blood pressure
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure (SBP) | Immediately after the intervention
  SBP mean difference and 95% CIs in mmHg
Diastolic Blood Pressure (DBP) | Immediately after the intervention
  DBP mean difference and 95% CIs in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: John L. Sievenpiper, MD,PhD,FRCPC, Principal Investigator — University of Toronto
Locations (1):
- Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no individual data collected. However, data from all included studies will be published in the manuscript and supplementary material